CLINICAL TRIAL: NCT00711347
Title: Intraoperative Floppy Iris Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Rick Potvin, Alcon Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M07-013
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2010-08

CONDITIONS: Cataract; Floppy Iris Syndrome
Keywords: Discovisc; Ophthalmic Visco Surgical Device
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- DisCoVisc (Active Comparator): Alcon's DisCoVisc Ophthalmic Viscosurgical Device (OVD) used at time of cataract surgery
  Interventions: Device: DisCoVisc
- Healon5 (Active Comparator): Abbott Medical Optic's (AMO) Healon5 Ophthalmic Viscosurgical Device (OVD) used at time of cataract surgery
  Interventions: Device: Healon5

INTERVENTIONS:
Device: DisCoVisc — Use of Alcon's DisCoVisc Ophthalmic Viscosurgical Device(4% sodium chondroitin sulfate, 1.65% sodium hyaluronate) during cataract surgery with intraocular lens implantation.
  Arms: DisCoVisc
Device: Healon5 — Use of Abbott Medical Optics (AMO) Healon5 Ophthalmic Viscosurgical Device (2.3% Sodium Hyaluronate) during cataract surgery with intraocular lens implantation.
  Arms: Healon5

SUMMARY:
An assessment of the surgical performance of DisCoVisc compared to Healon5 during cataract surgery with intraocular lens implantation where miotic/small pupils or intraoperative Floppy Iris Syndrome exists.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with floppy iris syndrome
* operable bilateral cataracts

Exclusion Criteria:

* Intraocular Pressure (IOP) > 21mmHg
* ocular inflammatory disease
* systemic or ocular diseases affecting Endothelial Cell Count

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Contact Alcon Call Center for Study Locations, Fort Worth, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were scheduled for routine, primary, bilateral cataract extraction with subsequent insertion of an intraocular lens implant and demonstrating miotic/small pupils or intraoperative floppy iris syndrome. Additionally patients were free of ocular co-morbidities that may affect results.
Pre-assignment Details: During the preoperative exam, subjects were examined to ensure they met the inclusion/exclusion criteria. Only subjects who signed an informed consent and qualified to be in the study by meeting all inclusion/exclusion criteria were enrolled. Patients were randomized (Excel based schedule) based on enrollment order.
Groups:
- DisCoVisc: Alcon's DisCoVisc used at time of surgery
- Healon5: Abbot Medical Optics (AMO) Healon5 used at time of surgery
Period: Overall Study
Arm/Group | DisCoVisc | Healon5
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DisCoVisc | Healon5 | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 13 | 13 | 26
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Corneal Endothelial Cell Loss
Description: Endothelial cell loss/gain is measured by comparing the preoperative assessment of endothelial cell density against postoperative measurements. Measurements are made with a specular microscope, which takes a picture and numbers endothelial cells. This endpoint compares the assessment done at 1 month against the assessment done at baseline. A negative number indicates a loss of endothelial cells, a positive number indicates a gain in endothelial cells.
Time Frame: 1 month
Population: 14 patients/28 eyes in each group.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | DisCoVisc | Healon5
Number analyzed (Participants) | 14 | 14
Percent change | 9.85 (14.07) | -3.68 (16.52)

2. Secondary Outcome: Intraocular Pressure (IOP)
Description: Intraocular Pressure (IOP) is assessed with a slit lamp by means of Applanation (Goldmann) tonometry. This type of tonometry uses a small probe to gently flatten part of your cornea to measure eye pressure. The pressure in your eye is measured by how much force is needed to flatten your cornea, and measured in millimeters of mercury (mmHg). Normally, IOP should be less than 21 mmHg.
Time Frame: 1 Day Postoperative
Population: 14 patients/28 eyes in each group.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | DisCoVisc | Healon5
Number analyzed (Participants) | 14 | 14
mmHg | 16.93 (3.67) | 20.29 (11.19)

3. Secondary Outcome: Aqueous Signs - Cells
Description: Aqueous Cells are the foggy appearance given by protein that has leaked from inflamed blood vessels. This is evaluated by the surgeon one day post surgery and rated on the following scale: None, 0: 1-5 cells, 1: 6-15 cells, 2: 16-30 cells, 3: >30 cells
Time Frame: 1 Day Postoperative
Population: 14 patients/28 eyes in each group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DisCoVisc | Healon5
Number analyzed (Participants) | 14 | 14
Units on a scale | 0.93 (1.00) | 1.14 (0.95)

4. Secondary Outcome: Aqueous Signs - Flare
Description: Aqueous Flare refers to individual inflammatory cells. Aqueous flare is evaluated by the surgeon one day after surgery and rated on the following scale:
  0:No-Visible flare when compared with the normal eye.
  1. Mild-Flare visible against dark papillary background but not visible against iris background.
  2. Moderate-flare is visible with the slit-lamp beam aimed onto the iris surface as well as the dark papillary background.
  3. Severe-Very dense flare. May also present as a hazy appearance of anterior segment structures when viewed with low power magnification of the slit-lamp.
Time Frame: 1 Day Postoperative
Population: 14 patients/28 eyes in each group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DisCoVisc | Healon5
Number analyzed (Participants) | 14 | 14
Units on a scale | 0.43 (0.51) | 0.69 (0.48)

5. Secondary Outcome: Aqueous Signs - Edema
Description: Aqueous signs refers cornea edema evaluated by the surgeon one day after surgery. Corneal edema is evaluated by the following scale:
  0 = none
  1. = mild - slight localized or generalized edema
  2. = moderate - significant localized or generalized edema
  3. = severe - advanced localized or generalized edema
Time Frame: 1 Day Postoperative
Population: 14 patients/28 eyes in each group.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DisCoVisc | Healon5
Number analyzed (Participants) | 14 | 14
Units on a scale | 0.57 (0.65) | 0.79 (0.89)

6. Secondary Outcome: Surgeon Survey
Description: Survey completed by the surgeon to evaluate use of the product during surgery. Responses are rated on the following scale and the means of the responses are reported:
  Overall surgical difficulty: 1 - very easy; 2 - easy; 3 - neither easy nor difficult; 4 - difficult; 5 - very difficult
  Satisfaction with performance: 1 - strongly disagree; 2 - disagree; 3 - undecided/neutral; 4 - agree; 5 - strongly agree
  Ability to expand pupil: 1 - not effective; 2 - moderately effective; 3 - very effective
Time Frame: Time of Surgery
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DisCoVisc | Healon5
Number analyzed (Participants) | 14 | 14
Units on a scale
  Surgeon Survey: Overall Surgical Difficulty | 1.9 (0.8) | 2.5 (0.9)
  Surgeon Survey: Satisfaction with Performance | 4.6 (0.5) | 3.6 (1.0)
  Surgeon Survey: Ability to Expand Pupil | 2.9 (0.4) | 2.9 (0.3)

ADVERSE EVENTS:
Arm/Group | DisCoVisc | Healon5
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written agreement.